CLINICAL TRIAL: NCT03252028
Title: Rapid Test for Detection of the Focus of Infection in Post Neurosurgical Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fariba Nayeri (Other)
Responsible Party: Sponsor-Investigator, Fariba Nayeri, MD, PhD, associated professor, University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Other Study IDs: LINPEAS
Record Dates: First submitted 2017-08-13; First posted 2017-08-17 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Infection, Bacterial; Antibiotic Resistant Infection; Diagnostic Self Evaluation; Meningitis, Bacterial; Nosocomial Infection
Keywords: Hepatocyte growth factor, Nosocomial infections, VAP, Meningitis, In vitro, point of care, rapid test
MeSH Terms: conditions — Bacterial Infections; Meningitis, Bacterial; Cross Infection; Deafness, Autosomal Recessive 39; Meningitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples from CSF, Sputum, Urine, Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Due to anatomical restrictions, the inflammatory response to intra-cerebral bacterial infections exposes swollen brain tissues to pressure and ischemia, resulting in life-threatening damage. However, diagnosing meningitis in patients after neurosurgery is complicated, due to brain tissue damage and changes in cerebrospinal fluid (CSF) caused by surgery. Hepatocyte growth factor (HGF) is a local, acute-phase protein. Previous studies on community-acquired septic meningitis reported high levels of intrathecal-produced HGF.

Aim: The aim of present study is to evaluate a new platform for qualitative determination of HGF in body fluids and revealing the site of injury.

Method: Based on a reverse-methachromacy method, strips are prepared. The surface on the strip changes colour to blue upon contact with HGF.

Plan: CSF, urine and sputum of patients that develop fever post neurosurgery are analysed with the test and the results compared with conventional diagnostic methods.

Clinical value: A rapid, equipment-free test gives the opportunity to identify the infectious focus in the infected organ long before culture results are available.

DETAILED DESCRIPTION:
Hepatocyte growth factor (HGF) is local acute phase protein with regenerative properties that become biologic inactive during chronic inflammation and loses the binding affinity to glycosaminoglycan in the extracellular ma-trix. HGF is excreted into the gastrointestinal tract and is not detected in normal urine. Nosocomial meningitis can occur when brain surgical procedures are complicated by infection. Due to underlying CNS disease processes and CNS devices in situ, the principal agents of nosocomial bacterial meningitis differ from the agents of community-acquired meningitis. For example, in nosocomial infections, slow growing, opportunistic microorganisms predominate. The CSF leukocyte profile is affected by intracerebral haemorrhage, and CSF lactate might be elevated, due to ischemia. Moreover, altered consciousness can make it difficult to establish a diagnosis in patients on ventilators that develop fever after neurosurgical operations. In other words, it is often difficult to determine whether the injured brain has been invaded by environmental bacterial flora.

Due to the challenges in establishing a diagnosis, and the lack of gold standards, physicians are motivated to treat suspected infections in serious dis-eases with broad-spectrum antibiotics. The emerging problems of multiple-resistance bacteria, high costs, and complications related to new antibiotics have called for diagnostic tests that can minimize antibiotic consumption.

Currently, the diagnosis of bacterial meningitis remains based on standard methods of direct microscopy, differential analyses of white blood cells, lactate, and protein, and cultures of blood and CSF . However, post-neurosurgical infections are difficult to distinguish from the effects of neurosurgical procedures. Moreover, due to prophylaxis treatments, the cultures are negative in a large group of patients, and the presence of skin flora, like Coagulase negative Staphylococcus or Propionbacterium acnes, may indicate either infection or contamination. Survival from this life-threatening condition depends on a rapid diagnosis and prompt empirical antibiotic therapy designed to cover the likely pathogens.

Where is the focus of infection? Is it a bacterial (septic) meningitis? Is the broad-spectrum antibiotic administration indicated? The background of the project: An invasion of bacteria into the central nervous system (CNS) is followed by a rapidly evolving inflammatory process that affects the arachnoid space, the pia mater, and the cerebrospinal fluid (CSF). This condition leads to clinical symptoms of headache, fever, and meningism. The inflammatory response is caused by the release of various pro-inflammatory cytokines from meningeal cells into the subarachnoid space. As a result, neutrophils move into the subarachnoid space and cause pleocytosis in the CSF. The consequences include the breakdown of the blood-brain barrier, cerebral oedema, reduced cerebral blood flow, focal areas of hypo perfusion, vascular thrombosis, ischemia, enhanced glucose metabolism via the anaerobic glycolytic pathway, and enhanced lactate accumulation in the brain and CSF [1]. Survival from this life-threatening condition depends on a rapid diagnosis and prompt empirical antibiotic therapy designed to cover the likely pathogens.

Other causes of febrile meningitis include acute viral meningitis and non-pyogenic meningitis, where the clinical picture is typically sub-acute or chronic. The diagnostic procedures consist of a lumbar puncture to analyse the CSF for cells and bacteria, microbiological cultures of blood and CSF, serological tests involving PCR and antigen-detection, and radiographic techniques [2]. In community-acquired meningitis, a combination of discriminating values from the CSF analysis can differentiate acute bacterial meningitis from other, non-ambulatory causes with quite high sensitivity [3].

Nosocomial meningitis can occur when brain surgical procedures are complicated by infection [2]. Due to underlying CNS disease processes and CNS devices in situ, the principal agents of nosocomial bacterial meningitis differ from the agents of community-acquired meningitis. The CSF leukocyte profile is affected by intra-cerebral haemorrhage, and CSF lactate might be elevated, due to ischemia. Moreover, altered consciousness can make it difficult to establish a diagnosis in patients on ventilators that develop fever after neurosurgical operations.

Hepatocyte growth factor (HGF) is produced by mesenchymal cells during organ injury. It is produced as a single-chain precursor protein, and it is activated at the site of injury by proteolysis cleavage, resulting in a double-chained active form of HGF [4]. Active HGF stimulates cell division [4] and cell motility, and it promotes normal morphogenic structure [5] in epithelial cells adjacent to injured areas. Thus, HGF induces regeneration and re-pair of damaged tissue [6]. High levels of systemic HGF have been detected during injuries caused by infection [7]. In bacterial meningitis, pneumonia and acute bacterial gastroenteritis, there is local production of HGF at the site of infection [7-9]. HGF produced locally during bacterial infection is biologically active [10]. Application of biologically active HGF promoted healing of chronic leg ulcers in a pilot study [11]. Effective antibiotic therapy reduces systemic HGF levels during infection [12-13]. HGF might be regarded as a local acute phase protein with healing properties [14].

The quality of endogenous HGF binding to receptors can be assessed with surface plasmon resonance (SPR), an optical technique appropriate for clinical studies that can determine the affinity of a protein for several ligands [15]. SPR-based assessment of HGF binding affinity for its receptors, c-Met and heparan sulphate proteoglycan (HSPG), could rapidly and sensitively distinguish HGF variants with different biological activities [16-17].

We have previously studied the concentration of HGF in CSF for patients with community- acquired meningitis [7]. We have also shown that the presence of biologically active HGF at the site of injury indicates an acute local inflammation [18]. During a recent study we have assessed whether HGF concentrations and HGF binding affinity for its receptors might serve as markers to distinguish between meningitis associated with neurosurgery and other causes of infection. We determined the concentration and binding affinity of HGF in patients with either community-acquired meningitis or neurosurgery-associated meningitis, and compared the results to either patients with Alzheimer's disease or controls with normal CSF. We have shown that determination of HGF in CSF might be used as an indicator, complementary to clinical status and routine laboratory findings, for diagnosing bacterial invasion into the CSF at an early stage of disease [18].

The problem:

Case report: 76 years old woman with high blood pressure was found by her neighbours, unconscious in her garden 28th October 2009. The CT scan revealed subarachnoid haemorrhage and neuro-angiography revealed 3 aneurysms. She was admitted to the Department of neurosurgery and operated 29th October with ventricular drainage and endovascular occlusion of the aneurysms. She was extubated post-surgery however she suffered from left arm and leg paralysis and tiredness. Since 30th October she had low grade of fever and slightly increased CRP and procalcitonin. Cerebrospinal fluid showed 170.000 red and 630 white blood cells and lactate 5.8. The chest X-ray showed a suspect infiltration. The blood and CSF cultures were secured. The cultures taken from 5th November revealed significant growth of Enterobacter cloacae and Staphylococcus aurous in urine and growth of Staphylococcus aurous in the nasopharynx. She received no antibiotic therapy and the parameters decreased spontaneously but low grade of fever continued. The CSF blood cells increased to 23000 red and 106 white blood cells (11th November), and CSF lactate was 4.5 (lumbar drainage). Although CRP was in the normal range she received meropenen 2g x 3 under suspicion bacterial meningitis. First on 19th November the CSF cultures taken on 11th November revealed growth of Propionibacterium acnes. The antibiotic regime continued until 23th November. She suffered from disorientation, fatigue, and had hydrocephalus. She underwent shunt operation 23th November. She died 2nd December 2009. High concentration of HGF and elevated binding affinity to HSPG was found in CSF analysis already 2nd November.

Due to the challenges in establishing a diagnosis, and the lack of gold standards, physicians are motivated to treat suspected infections individually because there is no diagnostic method that can identify the infections focus in time. PCR for bacterial panel and virus detection in CSF is sensitive method. However it might detect the colonized bacteria as well. The presence of bacteria is not the same as infection. Therefore in cases of bacterial meningitis especially post brain surgery and the foreign bodies that are inserted in the brain we cannot rely on positive or negative cultures totally. A complementary method (for the standard available methods at laboratory) with high negative predictive value increases the specificity of tests and decreases the costs, time and complications such as hospital acquired infections (HAI) profoundly.

The Method, Reverse Methachromacy:

The N-terminus of HGF (Hairpin Loop) has been identified as the binding site to both c-Met and HSPG. There is a high correlation between binding of HGF to HSPG and to dextran sulphate in SPR system (fig 1). Metochromasia is a characteristic colour change that certain aniline dyes exhibit when bound to chromo trope substances [19].This phenomenon has been widely used in the study of tissue sections. Methylene blue (O-toluidine) is considered an excellent metachromatic dye. Upon binding to high molecular weight polysaccharides, such as dextran sulphate, the colour of the indicator solution changes from blue to red [19].

Combinations of dextran sulphate and O-toluidine in different proportions produce purple-red coloured solutions of varying intensity. Coated customized filter papers make up surfaces that are placed on strips. When in con-tact with biological solutions, the sample HGF competitively replaces O-toluidine for binding to dextran sulphate and the colour of the surface returns to blue (Fig 2). This platform detects the presence of HSPG-binding proteins such as HGF in body fluids including expectorant, urine, ulcer secretions, cerebrospinal fluid, and joint effusion during infection. High amounts of protein or high pH do not cause non-specific reactions with this device.

The study plan:

Study leader: Amir Ramezani

The Procedure:

CSF specimens, urine and sputum (n=500) are collected from patients (1-99 years old) that have undergone brain tumour surgery, intracerebral haemorrhage, shunt dysfunction or skull fracture. The specimens are kept frozen in -20° C until analyses were performed. There are no exclusion's criteria.

Controls Alzheimer's disease (n=20)

* CSF samples were collected and kept frozen from patients (N=20) that were diagnosed with Alzheimer's disease at the Memory Clinic, Skåne University Hospital in Malmö. The revised DSM-III and NINDS-ADRDA criteria were used for diagnosis of Alzheimer's dementia (this study group has been included in previous study).
* Normal CSF
* This group consists of patients who have undergone lumbar puncture to rule out meningitis, and they had normal CSF.
* Analysis of ligand-binding affinity with surface plasmon resonance
* The biological activity of HGF is analysed with SPR. We measure the binding affinity to HSPG (Sigma-Aldrich, St. Louis, MO, USA) and to a c-Met recombinant chimera (R&D Systems), as previously described.
* Measurements of HGF concentrations in samples A specific enzyme-linked immunosorbent assay (ELISA) kit (Quantikine Human HGF immunoassay, minimum detectable limit: 0.04 ng/mL; R&D Systems, Minneapolis, MN, USA) was used to determine HGF concentrations in CSF, sputum and urine according to the manufacturer's instructions. All measurements were performed with an ELISA reader (Expert96; AsysHitech GmbH, Eugendorf, Austria) at 450 nm, which was calibrated with the recombinant human HGF reference samples and the standards provided in the kit.
* Reverse methachromacy The study strip test is performed on all specimens.
* Routine laboratory assessments
* CSF is analysed to determine parameter values at the Departments of Clinical Chemistry, University Hospitals, in Linköping. All cultures, PCR assays, antigen detection assays, and serological assessments are performed at the Department of Microbiology, University Hospital, Linköping, Sweden.
* CSF-cells: Performed by manual phase contrast microscopy (Zeiss) using Jessen Chamber for counting the number of erythrocytes and leukocytes (polymorphonuclear neutrophils and monocytes).
* CSF lactate: Performed using benchtop blood gas analyzer ABL 800 (Radiometer Medical ApS Denmark).
* Antigen detection: Antigen (Streptococcus pneumonia, Haemophilus influenza, Neisseria meningitides group A, group B/Escherichia coli K1, group C and group Y/135, Streptococcus agalactiae) is detected by latex agglutination method Pastorex Meningitis™ (Bio-Rad, France).
* CSF culture: Performed in aerobe and anaerobe flasks as well as in Hematin plates.
* Virus detection PCR: Herpes virus type 1 and 2 (HSV1, HSV 2) and HZV DNA were detected by PCR. Human enterovirus (HEV) was analysed by automated instrument (Cepheid GeneXpert).
* Statistical analysis
* Because the HGF concentrations and binding affinity data are not normally distributed, non parametric tests Kruskal-Wallis test followed by the Mann-Whitney U test or the Wilcoxon matched pairs test are appropriate for analysis. The analysis of test performance shall be performed manually.

Clinical Evaluation of the Platform in a Dextran Sulphate-Containing Gel Using reverse methachromacy approach we have studied a total of 656 faeces samples with The sensitivity, specificity, positive predictive value, and negative predictive value as well as the accuracy were calculated in the following groups: verified infectious gastroenteritis (n=207) and other causes of diarrhoea, including IBD (n=268). The test could distinguish acute infectious gastroenteritis with a sensitivity of 96.6% and specificity 92.4%, and a positive predictive value of 90.9% and negative predictive value of 97.2%. The accuracy of test was 94.3%. No significant correlation between the test results and faeces calprotectin were found (R2=0·056). No significant correlation was observed between the results of the index test and the presence of blood in the faeces (R2=0·08) [20].

Clinical evaluation of HGF as a marker to distinguish septic meningitis from other causes of pleocytosis [18] The community-acquired septic meningitis showed significantly higher HGF concentration (p=0.0133), as well as HGF binding affinity to the c-Met and HSPG receptors (p=0.0007 and p=0.0009, respectively) compared to nosocomial meningitis. CSF samples from patients with septic meningitis (including both community-acquired and nosocomial) was significantly higher in HGF concentrations (p=0.0014), HGF binding to HSPG (p<0.0001), and HGF binding to c-Met (p<0.0001) compared to samples from patients with aseptic (viral and sub acute) meningitis. CSF samples from patients with septic meningitis was higher from samples from the control group (patients with normal CSF) and from patients with Alzheimer's disease in HGF concentration (p<0.0001, p=0.0010, respectively), HGF binding to HSPG (p<0.0001 and p=0.9, respectively), and HGF binding to c-Met (both p<0.0001).

Compared to samples from patients that had undergone neurosurgery and had other infectious diseases, CSF samples from patients with nosocomial meningitis had significantly higher HGF concentrations (p<0.0001) and HGF binding affinity to c-Met (p<0.0001) and HSPG (p=0.043) receptors (Figure 3-4).

Figure Legends Fig. 1. Sequence of part of the HGF α-chain. The enlarged codons code for amino acids important for binding to HSPG and the c-Met receptor.

Fig. 2. The theoretical support for the second approach for a device to de-tect the presence of HGF in body fluids during an infection. (1) Glucosaminoglycan (GAG) polymer chain with negative charges. (2) Positive TBO molecules attach to the polymer chain then are concentrated and form stacks. The colour changes from blue to red. (3) A sample with HGF is added, which binds to GAG. (4) TBO molecule stacks are destroyed and become freely dissolved TBO molecules. The colour changes from red to blue.

Figure 3: Flow chart of the selection of CSF specimens from patient and control groups. Extra samples are the samples taken during stay on ward from patients with nosocomial meningitis.

Figure 4: Properties of HGF derived from different CSF samples were analysed by using surface plasmon and ELISA techniques. (A) Binding to c-Met receptors; (B) Binding to HSPG receptors; (C) HGF concentrations (median). *p<0.05, **p<0.01, ***p<0.001, ****p<0.0001.

The rapid evolution and spread of antimicrobial-resistant bacteria in parallel with insufficient development of new active drugs seriously affect future anti-infective therapy of bacterial infections, especially those due to Gram-negative rods. Experts in the field estimate that by the next decade the world will have witnessed the wide dissemination of untreatable (or next-to untreatable) infections, both within and beyond hospitals. To avoid or at least attempt to retard this crisis, many researchers have dedicated their efforts to elucidate factors favouring the emergence and global spread of antimicrobial resistant bacteria. An effective strategy to limit the emergence of multiple resistant strains might include directing the antibiotic therapy by identifying cases that should or should not be treated with antibiotics, avoiding wide-spectrum antibiotic administration, and promoting more specific treatments.

What is needed is a simple, accurate, cost-effective and feasible test that answers to crucial questions.

In order to assess the clinical relevance and the performance of such a test there is not a better environment than the Swedish healthcare that provides the relevant and modern assessment of diseases and evidence-based therapy for nearly all patients. Such an environment is an opportunity to perform the patient inclusion and evaluation of the study test in comparison to the most reliable standard tools such as cultures, blood tests and X-rays. These resources are not available automatically in any other centre with such reliable, non-commercial and impartial properties.

dnr 2015-429-32

ELIGIBILITY:
Inclusion Criteria:

* all post neurosurgical patients with suspect infection or fever

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all post-neurosurgical patients in neuro intensive care unit university hospital Linkoping, Sweden
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-12-02 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
detection of infections in intensive care unit | 4 years
  analyse of different body fluids to detect the focus of infections post neurosurgical fever

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Neurosurgery dept. University Hospital, Linköping, Östergötland County
  - Neurosurgery department, University Hospital, Linköping, Östergötland County